CLINICAL TRIAL: NCT02097524
Title: Single-dose Study to Describe the Pharmacodynamics (PD) and Safety of Sarilumab (REGN88/SAR153191) and Tocilizumab in Adults With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6R88-RA-1309
Record Dates: First submitted 2014-03-03; First posted 2014-03-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sarilumab - dose 1 (Experimental): Single subcutaneous (SC) injection of Sarilumab, dose 1, plus methotrexate background treatment (dispensed and dosed according to local practice)
  Interventions: Drug: Sarilumab
- Sarilumab - dose 2 (Experimental): Single SC injection of Sarilumab, dose 2, plus methotrexate background treatment (dispensed and dosed according to local practice)
  Interventions: Drug: Sarilumab
- Tocilizumab - dose 1 (Active Comparator): Single intravenous (IV) administration of Tocilizumab, dose 1, plus methotrexate background treatment (dispensed and dosed according to local practice)
  Interventions: Drug: Tocilizumab
- Tocilizumab - dose 2 (Active Comparator): Single IV administration of Tocilizumab, dose 2, plus methotrexate background treatment (dispensed and dosed according to local practice)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Sarilumab
  Other Names: REGN88; SAR153191
  Arms: Sarilumab - dose 1; Sarilumab - dose 2
Drug: Tocilizumab
  Arms: Tocilizumab - dose 1; Tocilizumab - dose 2

SUMMARY:
The main purposes of this study are to describe the pharmacodynamic effects, safety and pharmacokinetics of a single dose of sarilumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RA as defined by the 2010 revised American College of Rheumatology (ACR)
2. ACR Class I-III functional status, based on the 1991 revised criteria
3. Treated for a minimum of 12 weeks with Methotrexate with a stable dose of MTX for at least 8 weeks prior to screening visit

Exclusion Criteria:

1. Patients less than 18 years of age or minimum legal age
2. Prior treatment with any biologic anti-Interleukin 6 (IL-6) or IL-6 Receptor (IL-6R) antagonists
3. Use of parenteral corticosteroids or intra-articular corticosteroids within 4 weeks prior to screening
4. Use of oral corticosteroids in a dose higher than prednisone 10 mg or equivalent per day, or a change in dosage within 4 weeks prior to randomization
5. Participation in any clinical research study that evaluated an investigational drug or therapy within 5 half-lives or 60 days of the screening visit, whichever is longer
6. Treatment with oral/ biologic DMARDs (disease-modifying antirheumatic drugs), other than MTX, within a certain amount of time prior to screening visit
7. Active or suspected TB or at high risk of contracting TB
8. Fever, or chronic, persistent, or recurring infections requiring active treatment
9. HIV positive

Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial therefore not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
PD parameters | baseline through week 4
  Pharmacodynamic (PD) parameters, what a drug does to the body, will be collected from baseline through week 4:
  * the time to nadir (or peak)
  * change from baseline
  * area under the curve (AUC)

SECONDARY OUTCOMES:
Percentage of TEAEs | baseline through week 6
  Percentage of patients with treatment-emergent adverse events (TEAEs) from baseline through end of study (week 6).
PK parameters | baseline through week 4
  Pharmacokinetic (PK) parameters, what the body does to a drug, will be collected from baseline through week 4:
  * AUC
  * CL (clearance)
  * Cmax (the peak concentration)
  * t1/2 (observed terminal half-life)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Orange, California
  - DeLand, Florida
  - Edgewater, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Granger, Indiana
  - Grand Blanc, Michigan
  - Charlotte, North Carolina
  - Cinicinnati, Ohio
  - Memphis, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Channelview, Texas
  - Dallas, Texas
  - Houston, Texas
  - Mesquite, Texas
  - Plano, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Kovalenko P, Paccaly A, Boyapati A, Xu C, St John G, Nivens MC, Davis JD, Rippley R, DiCioccio AT. Population Pharmacodynamic Model of Neutrophil Margination and Tolerance to Describe Effect of Sarilumab on Absolute Neutrophil Count in Patients with Rheumatoid Arthritis. CPT Pharmacometrics Syst Pharmacol. 2020 Jul;9(7):405-416. doi: 10.1002/psp4.12534. Epub 2020 Jun 20. PMID 32453485
- [Derived] Emery P, Rondon J, Parrino J, Lin Y, Pena-Rossi C, van Hoogstraten H, Graham NMH, Liu N, Paccaly A, Wu R, Spindler A. Safety and tolerability of subcutaneous sarilumab and intravenous tocilizumab in patients with rheumatoid arthritis. Rheumatology (Oxford). 2019 May 1;58(5):849-858. doi: 10.1093/rheumatology/key361. PMID 30590833